CLINICAL TRIAL: NCT06191536
Title: The Effect of PVE Applied in Addition to Pilates on Premenstrual Symptoms, Pain, Sleep and QoL in Individuals With Premenstrual Syndrome
Brief Title: The Effect of PVE Applied in Addition to Pilates on Premenstrual Symptoms, Pain, Sleep and QoL in Individuals With PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, osman coban, Asst. Professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UskudarUniversitesi
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Premenstrual Syndrome; Pelvic Floor Disorders; Quality of Life
Keywords: Premenstrual Syndrome; Pelvic Floor Exercises; Pilates; Quality of Life; Pain
MeSH Terms: conditions — Premenstrual Syndrome; Pelvic Floor Disorders; Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Group (PG) (Experimental): Pilates exercises will be performed under the supervision of a certified pilates instructor.
  Pilates exercises will be performed for 50 minutes, 2 days a week for 8 weeks.
  Interventions: Other: Pilates
- Pelvic Floor Exercise Group (PFEG) (Active Comparator): It consists of voluntary pelvic floor muscle contractions applied in addition to pilates exercises.
  Pelvic floor muscle contractions involve maximum contraction of the pelvic floor muscles alternately for five repetitions during exhalation.
  Pelvic floor exercises will be applied under the supervision of a pelvic floor certified physiotherapist.
  In addition to pilates exercises, pelvic floor exercises will be applied 2 days a week, 50 minutes, for 8 weeks.
  Interventions: Other: Pilates; Other: Pelvic floor exercises

INTERVENTIONS:
Other: Pilates
Other: Pelvic floor exercises
  Arms: Pelvic Floor Exercise Group (PFEG)

SUMMARY:
Premenstrual syndrome (PMS) is a condition that occurs with physical and psychological symptoms in the late luteal phase of the menstrual cycle in women and affects the physical and mental well-being of the individual. Physiological symptoms; edema, headache, fatigue, weight gain and breast swelling and tenderness, and psychological symptoms; It can be seen as tension, anger, depressed mood or stress. Although it usually ends with the onset of menstruation, its repetition with each menstrual cycle affects the individual's pain coping strategies, sleep and quality of life.

Different methods such as pharmacological agents, physiotherapy applications, nutrition and lifestyle adjustments, breathing exercises, stress management, meditation and cognitive behavioral therapy are used to cope with PMS, which appears with symptoms of different severities from individual to individual.

DETAILED DESCRIPTION:
Exercise; It is known to have positive physical and psychological effects on PMS symptoms by reducing muscle cramps, increasing circulation and controlling the neuromuscular system. Pilates, as an exercise method that combines body-mind conditioning with breathing control and focuses on lumbopelvic stability and targets core stabilization, is also thought to have a significant effect on increasing pelvic floor muscle strength by performing it together with pelvic floor muscle contraction. In addition, considering the anatomical connection of the pelvic floor muscles with other core muscles, it has been observed that pelvic floor muscle contractions also occur during abdominal muscle contraction. The pelvic floor consists of a group of muscles and connective tissues that extend like a sling across the pelvic floor; It consists of two layers, the superficial perineal muscles and the deep pelvic diaphragm, and provides support to the pelvic organs, bladder and elements of the spine. Pelvic floor exercises are a safe and effective means of decreasing the symptoms and signs of pelvic disorders. In the literature, it is seen that these exercises are effective in urinary incontinence.

There is no study examining the effect of pelvic floor muscle training combined with pilates on PMS symptoms. The purpose of this study; To examine the effects of pelvic floor exercises, in addition to pilates exercises, on PMS symptoms, pain, sleep and quality of life in individuals with premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to participate in research
* Getting a score of 111 or higher on the PMS Scale,
* Experiencing premenstrual symptoms for at least 3 months,
* Having a pain score of at least 4 on the Visual Analogue Scale during any menstrual period within the last 3 months.
* Regular menstrual cycle for 12 months (24-35 days),

Exclusion Criteria:

* Being under 18 years of age,
* Change in menstrual characteristics after PMS diagnosis,
* Having a chronic or physical illness that prevents you from doing Pilates.
* People who have had surgery in the last 6 months,
* Individuals with musculoskeletal system problems,
* Individuals with chronic diseases,
* People receiving hormone therapy,
* Pregnant individuals,
* People with urinary, genital or gastrointestinal disorders,
* People who have had hysterectomy surgery.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | 6 months
  The Premenstrual Syndrome Scale (PMSS) is a 44-item questionnaire based on a five-point Likert-type scale with scores ranging from 1 to 5. (Never, Rarely, Sometimes, Often, Constantly) Pmss has nine subscales, including Depressive Affects, Anxiety, Fatigue, Irritability, Depressive Thoughts, Pain, Appetite Changes, Sleep Changes, and Swelling. The PMSS total score is the sum of the scores of these nine subscales. The lowest score that can be obtained from the scale is 44 and the highest score is 220. The higher the score, the greater the intensity of PMS symptoms. In order to be diagnosed with PMS, it is necessary to get 50% of the total score (111 points).

SECONDARY OUTCOMES:
SF-12 | 6 Months
  Similar to SF-36, SF-12 includes physical functionality (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functionality (1 item). It consists of 8 subscales and 12 items, including emotional role (2 items) and mental health (2 items). While items related to physical and emotional roles are answered as dikatomis (yes or no), other items have Likert-type options ranging from 3 to 6. It is possible to obtain separate scores for each subscale, the score of the subscales varies between 0 and 100, with a higher score representing better health.
Pittsburgh Sleep Qualıty Index (PUKI) | 6 months
  PSQI is a sleep questionnaire that helps evaluate the person's sleep quality, amount of sleep, and the presence and severity of sleep disorders for the last month.
  This scale has 19 items and measures seven subcomponents of sleep quality, including subjective sleep quality, time to fall asleep, sleep duration, habitual sleep efficiency, sleep disturbances, sleeping pill use, and daytime dysfunction. The total PSQI score is obtained by summing the seven subscores and the total score is between 0-21. Each component is evaluated on a scale of 0-3 points. PSQI total score clearly distinguishes good sleepers (PSQI total score ≤5) from poor sleepers (PSQI >5).
Visual Analogue Scale (VAS) | 6 Months
  Visual Analogue Scale (VAS) is an evaluation method used to convert the pain perception level, which cannot be measured numerically, into a numerical form. In the evaluation, two extreme definitions of pain were written at both ends of a 100 mm line (I have no pain at one end, the most unbearable pain at the other end). The patient was asked to indicate where his/her current situation corresponds to on this line by drawing a line, placing a dot, or pointing. The distance from the point where there was no pain to the point marked by the patient, measured in mm with a ruler, showed the patient's pain level. Pain level was recorded as activity and rest VAS in the absence of bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: osman coban, PhD, Principal Investigator — Uskudar University
Locations (1):
- Heracity Pilates, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results of the study will be shared.

REFERENCES:
- [Background] Culligan PJ, Scherer J, Dyer K, Priestley JL, Guingon-White G, Delvecchio D, Vangeli M. A randomized clinical trial comparing pelvic floor muscle training to a Pilates exercise program for improving pelvic muscle strength. Int Urogynecol J. 2010 Apr;21(4):401-8. doi: 10.1007/s00192-009-1046-z. Epub 2010 Jan 22. PMID 20094704
- [Background] Leite A, Matignon A, Marlot L, Coelho A, Lopes S, Brochado G. The Impact of Clinical Pilates Exercises on Tension-Type Headaches: A Case Series. Behav Sci (Basel). 2023 Jan 27;13(2):105. doi: 10.3390/bs13020105. PMID 36829334
- [Background] Yaray O, Akesen B, Ocaklioglu G, Aydinli U. Validation of the Turkish version of the visual analog scale spine score in patients with spinal fractures. Acta Orthop Traumatol Turc. 2011;45(5):353-8. doi: 10.3944/AOTT.2011.2528. PMID 22033000
- [Background] Soylu C, Kutuk B. Reliability and Validity of the Turkish Version of SF-12 Health Survey. Turk Psikiyatri Derg. 2022 Summer;33(2):108-117. doi: 10.5080/u25700. English, Turkish. PMID 35730511